CLINICAL TRIAL: NCT00987506
Title: Evaluation of a XIENCE V® Endoprothesis Used for Coronary Angioplasty, for LPPR (List of Reimbursable Products and Services) Indications in Patients Monitored for 2 Years in France
Acronym: Far XIENCE V®
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: F330702
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Disease
Keywords: drug eluting stents; Stents; Angioplasty; Chronic coronary occlusion; Stent thrombosis; Vascular disease; Myocardial ischemia; Coronary artery stenosis; Coronary Disease; Coronary Artery Disease; Coronary Restenosis
MeSH Terms: conditions — Coronary Artery Disease; Vascular Diseases; Myocardial Ischemia; Coronary Stenosis; Coronary Disease; Coronary Restenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- XIENCE V®: Participants receiving XIENCE V® EESS
  Interventions: Device: XIENCE V®

INTERVENTIONS:
Device: XIENCE V® — Participants with placement of a XIENCE V® EESS

SUMMARY:
The objective of this study is to prepare elements of response to the Haute Autorité de Santé (High Health Authority) of France, which is expecting data relating to the routine use of XIENCE V® endoprothesis within the 5 years following its marketing.

ELIGIBILITY:
Inclusion Criteria:

All patients enrolled in the study must :

* be at least 18;
* be covered by Social Security
* agree to be enrolled in the study (sign the informed consent after reading the information letter).

In addition, the Xience V endoprothesis implantation must be performed following the LPPR indications here under :

Treatment of coronary heart disease attributable to de novo lesions (reference vessel with a 2.5 to 3.5 mm) of native coronary arteries, solely in the following groups of patients :

* patients with diabetes ;
* lesions of small vessels (diameter < 3 mm);
* long lesions (longer than 15 mm) ;
* stenosis of proximal anterior intraventricular septum .

The use of the Xience V stent is limited to one per patient, except :

* in case of acute occlusive dissection where three stents, maximum, may be covered ;
* for the pluritroncular diabetic patient, in case a bypass is contra-indicated : a stent per artery, with a limit of three per patient, may be covered.

Exclusion Criteria:

* Pregnant women
* Patients with:

  * a non cardiac vital prognosis endangered during the year following the implantation ;
  * less than 72 hours myocardial infarction ;
  * lower left ventricular ejection fraction < 30 % ;
  * an allergy to the platelets antiaggregant treatment, to heparin, chrome cobalt alloy, or to the angiography contrast medium ;
  * a stenosis of the unprotected common trunk;
  * a lesion with calcifications that cannot be pre-dilated;
  * a thrombus that can be detected by angiography on the lesion to be treated ;
  * an intra-stent re-stenosis.

Are also excluded :

* patients having had an angioplasty with implantation of an endoprothesis on the same vessel;
* patients having had an angioplasty with implantation of an endoprothesis during the 6 previous months ;
* Patients unable to keep a treatment associating aspirin and thiénopyridines for at least 6 months;
* Patients residing abroad or who cannot be monitored according to the modalities of the study ;
* Patients unable to give on their own free will their informed consent ; On the other hand, in absence of clinical validation, the other sub-groups of at risk patients (notably bifurcation lesions and pluritroncular lesions) cannot be considered , taken alone, as indications for the use of Xience V.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population Description * Definition: For observational studies only, a description of the population from which the groups or cohorts will be selected (e.g., primary care clinic, community sample, residents of a certain town).
Sampling Method: Non-Probability Sample
Enrollment: 1165 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Occurrence rate of new revascularisation (by a new angioplasty or coronary bypass) of the lesion(s) that had received the XIENCE V® endoprothesis, one year after its implantation. | 1 year

SECONDARY OUTCOMES:
Determine the occurrence rate of new revascularisation(s) after endoprothesis implantation | 18 and 24 months
Determine the occurrence rate of Major Cardiac Events | 6, 12, 18 and 24 months
Determine the occurrence rate of stent thrombosis as defined by the Academic Research Consortium | 6, 12, 18 and 24 months
The occurrence rate of death of cardiac origin | 6, 12, 18 and 24 months
Determine the occurrence rate of myocardial infarction | 6, 12, 18 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Didier Blanchard, MD, Principal Investigator — Hôpital Européen Georges-Pompidou
Locations (57):
- France (57):
  - Clinique De L'Europe, Amiens
  - CH Universitaire, Angers
  - Hopital Prive D'Antony, Antony
  - Clinique La Casamance - UCV, Aubagne
  - Clinique La Casamance-Vista, Aubagne
  - Clnique Rhone-Durance, Avignon
  - Clinique LaFourcade, Bayonne
  - CH Jean Minjoz, Besançon
  - Polyclinique Du Bois Bernard, Bois-Bernard
  - CH Jacques Coeur, Bourges
  - Hôpital de la Cavale Blanche-CHU, Brest
  - CH Prive Saint-Martin, Caen
  - Hopital Albert Schweitzer, Colmar
  - Clinique Des Cedres, Cornebarrieu
  - Polyclinique Louis Pasteur, Essey-lès-Nancy
  - Centre Cardiologique D'Evecquemont, Évecquemont
  - CH Saint Louis, La Rochelle
  - CH DE Lagny- Marne La Valee, Lagny-sur-Marne
  - CMC De Parly II, Le Chesnay
  - Polyclinique Du Bois, Lille
  - CH ST Joseph St. Luc, Lyon
  - Clinique Generale De Marignane, Marignane
  - Centre Cardio-Vasculaire Valmante, Marseille
  - CH Prive Beauregard, Marseille
  - Institut Hospitalier Jacques Cartier, Massy
  - Clinique Les Fontaines, Melun
  - Clinique Du Millenaire, Montpellier
  - Hopital Emile Muller, Mulhouse
  - NCN-Nouvelles Cliniques Nantaises, Nantes
  - Clinique Ambroise Pare, Neuilly-sur-Seine
  - Hopital Prive Les Franciscaines, Nîmes
  - Polyclinique les Fleurs, Ollioules
  - Institut Mutualiste Montsouris, Paris
  - Association Clinique Bizet, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Clinique Saint-Pierre, Perpignan
  - CH General Marechal Joffre, Perpignan
  - Clinicque St. Martin, Pessac
  - Polyclinique de Poitiers, Poitiers
  - Hopital Claude Gallien - ICPS, Quincy-sous-Sénart
  - Polyclinique St. Laurent, Rennes
  - Hopital Pontchaillou, Rennes
  - Hopital Charles Nicolle-CHU, Rouen
  - C.M.C.O De La Cote D'Opale, Saint Martin Les Boulogne
  - Centre Cardilogique du Nord, Saint-Denis
  - Clinique De L'Orangerie, Strasbourg
  - Hopital Foch, Suresnes
  - Clinique De L'Ormeau-CCV Des Pyrenees, Tarbes
  - Clinique Pasteur, Toulouse
  - Clinque Pasteur, Toulouse
  - Hopital De Rangueil - CHU, Toulouse
  - Clinique Saint Gatien, Tours
  - Centre Hospitalier De Valenciennes, Valenciennes
  - Polyclinique De Vauban, Valenciennes
  - Hopital de Brabois_CHU Nancy, Vandœuvre-lès-Nancy
  - CH Bretagne Atlantique, Vannes
  - Clinique Du Tonkin, Villeurbanne